CLINICAL TRIAL: NCT00060424
Title: Allogeneic Hematopoietic Stem Cell Transplantation With Nonmyeloablative Conditioning for Patients With Chronic Lymphocytic Leukemia - A Multi-center Trial
Brief Title: Fludarabine Phosphate and Total-Body Irradiation Before Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Maloney, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1711.00; NCI-2010-01276 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2011-01116; 1711.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: B-Cell Prolymphocytic Leukemia; Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; T-Cell Prolymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Leukemia, Prolymphocytic, T-Cell | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Mycophenolic Acid; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor, transplant, GVHD prophylaxis) (Experimental): NONMYELOABLATIVE CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and TBI on day 0. TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant on day 0. GVHD PROPHYLAXIS: Patients receive cyclosporine PO every 12 hours on days -3 to 180 with taper on day 56 and mycophenolate mofetil PO every 12 hours on days 0-27.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Procedure: Hematopoietic Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplant
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; stem cell transplantation
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplant
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This clinical trial studies how well giving fludarabine phosphate together with total-body irradiation (TBI) before donor peripheral blood stem cell transplant works in treating patients with chronic lymphocytic leukemia or small lymphocytic leukemia. Giving low doses of chemotherapy, such as fludarabine phosphate, and TBI before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. Giving chemotherapy before or after peripheral blood stem cell transplant also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before and after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether nonmyeloablative allogeneic hematopoietic stem cell transplantation (HSCT) from matched-related donors can improve the probability of survival 18 months after treatment for fludarabine (fludarabine phosphate)-refractory, fludarabine phosphate, cyclophosphamide, and rituximab (FCR)-failed, or del 17p chronic lymphocytic leukemia (CLL) beyond that observed in historical controls (30%).

SECONDARY OBJECTIVES:

I. To assess the rate of relapse with allogeneic HSCT using nonmyeloablative conditioning for patients with fludarabine-refractory, FCR-failed, or del 17p CLL compared with historical data on autologous HSCT.

II. To estimate the incidence of grade 2-4 acute graft-versus-host disease (GVHD) and chronic GVHD in patients with CLL treated with low-dose TBI, fludarabine, peripheral blood stem cell (PBSC) infusion and immunosuppression with cyclosporine and mycophenolate mofetil.

III. To characterize the rate and types of infections with this regimen.

IV. To estimate the rate of transplant-related mortality in the first 200 days.

OUTLINE:

NONMYELOABLATIVE CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and TBI on day 0.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant on day 0.

GVHD PROPHYLAXIS: Patients receive cyclosporine orally (PO) every 12 hours on days -3 to 180 with taper beginning on day 56 and mycophenolate mofetil PO every 12 hours on days 0-27.

After completion of study treatment, patients are followed up at 12 and 18 months and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CLL (or small lymphocytic lymphoma) or diagnosis of CLL that progresses to prolymphocytic leukemia (PLL), or T-cell CLL or PLL
* Patients with B-Cell CLL or PLL who have at least one of the following:
* Failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing fludarabine (or another nucleoside analog, e.g. cladribine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing fludarabine (or another nucleoside analog)
* Failed FCR combination chemotherapy at any time point
* Had de novo of acquired "17p deletion" cytogenetic abnormality; patients should have received induction chemotherapy but could be transplanted in first (1st) complete response (CR)
* Patient has a suitable human leukocyte antigen (HLA)-matched related donor who is willing to undergo leukapheresis initially for collection of PBSC and subsequently for collection of peripheral blood mononuclear cells (PBMC) with filgrastim (G-CSF) mobilization and willing to donate stem cells
* DONOR: Related donor who is HLA phenotypically or genotypically identical at the allele level at HLA-A, -B, -C, -DRB1, and -DQB1
* DONOR: Donor must consent to G-CSF administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)

Exclusion Criteria:

* Infection with human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV)-1, or HTLV-2
* Active central nervous system (CNS) involvement with CLL
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers)
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Pregnant or breastfeeding women
* Karnofsky score =< 70
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Cytotoxic agents for "cytoreduction" (with the exception of imatinib mesylate [Gleevec], cytokine therapy, hydroxyurea, chlorambucil or Rituxan) within three weeks of the initiation of conditioning
* Active bacterial or fungal infections unresponsive to medical therapy
* Cardiovascular: cardiac ejection fraction < 40%; patients with poorly controlled hypertension despite multiple antihypertensives
* Pulmonary: diffusing capacity of carbon monoxide (DLCO) < 40%, total lung capacity (TLC) < 40%, forced expiratory volume in one second (FEV1) < 40% and/or requiring continuous supplementary oxygen, or severe deficits in pulmonary function testing as defined by pulmonary consultant service
* Liver function abnormalities: patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dL, or symptomatic biliary disease
* DONOR: Age < 12 years
* DONOR: Identical twin
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to filgrastim (G-CSF)
* DONOR: Current serious systemic illness

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (3):
- United States (2):
  - Veterans Administration Center-Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
  Italy | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of patients surviving 18 months post-transplant.
Time Frame: At 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
Participants | 15

2. Secondary Outcome: Rate of Relapse
Description: Number of patients with relapsed disease post-transplant. Relapse/progression is defined as 1) Physical exam/Imaging studies (nodes, liver, and/or spleen) ≥50% increase or new, 2) circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, or 3) lymph node Biopsy Richter's transformation.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
Participants | 8

3. Secondary Outcome: Acute Grade II-IV GVHD and Chronic (Extensive) GVHD
Description: Number of patients who developed acute/chronic GVHD post-transplant. aGVHD Stages
  Skin:
  a maculopapular eruption involving < 25% BSA a maculopapular eruption involving 25 - 50% BSA generalized erythroderma generalized erythroderma with bullous formation and often with desquamation
  Liver:
  bilirubin 2.0 - 3.0 mg/100 mL bilirubin 3 - 5.9 mg/100 mL bilirubin 6 - 14.9 mg/100 mL bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 3 skin and/or stage 1 gut involvement and/or stage 1 liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: aGVHD: 100 days after transplant; cGVHD: 1 Year after transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
Participants
  Acute GVHD | 10
  Chronic extensive GVHD | 10

4. Secondary Outcome: Rate and Types of Infections
Description: Number of infections patients experienced, by infection type.
Time Frame: 18 months
Measure: Number; unit: infections
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
infections
  Viral | 27
  Fungal | 13
  Fever of unknown origin | 6
  Bacterial | 53
  Other | 5

5. Secondary Outcome: Transplant-related Mortality
Description: Defined as death before day +200 not related to progression of disease.
Time Frame: At 200 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
Participants | 2

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis)
Serious Adverse Events (participants affected / at risk) | 7/21
Other Adverse Events (participants affected / at risk) | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis) (N=21)
Death following progression of GVHD (Immune system disorders) | 1 (1)
Death following disease progression post transplant (Immune system disorders) | 2 (2)
Cardiac Arrhythmia and Seizure (Cardiac disorders) | 1 (1)
Death: Sepsis/Renal failure/ with history of GVHD (Renal and urinary disorders) | 1 (1)
Severe abnormal pain due to gut GVH (Gastrointestinal disorders) | 1 (1)
Acute Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Perforated sigmoid diverticulitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor, Transplant, GVHD Prophylaxis) (N=21)
Neutropenia (Blood and lymphatic system disorders) | 10 (10) — Grades 3, 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) — Grades 3, 4
Minimal hydronephosis (Renal and urinary disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Acute Pulmonary Embolism (Cardiac disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Increased creatinine (Renal and urinary disorders) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) — due to ifosfamide
Renal failure (Renal and urinary disorders) | 1 (1)
Tumor lysis syndrome (Blood and lymphatic system disorders) | 1 (1) — Uric acid level of 10.4 mg/dL.
Typhlitis & Bowel Perforation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes